CLINICAL TRIAL: NCT05820321
Title: Effects of Dietary Nitrate Intake on Physical Performance of Middle-aged Women: a Randomized Trial
Brief Title: Effects of Dietary Nitrate Intake on Physical Performance of Middle-aged Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cicero Jonas R Benjamim, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BEET-MS
Record Dates: First submitted 2023-01-27; First posted 2023-04-19 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Postmenopausal; Menorrhagia; Physical Inactivity; Motor Activity
MeSH Terms: conditions — Menorrhagia; Sedentary Behavior; Motor Activity | interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Beetroot juice NO3) (Active Comparator): 8-day supplementation with beetroot juice rich in NO3 (400mg) during 8 days.
  Interventions: Dietary Supplement: Beetroot juice rich in nitrate
- Placebo (Beetroot juice without NO3) (Placebo Comparator): 8-day supplementation with beetroot juice NO3 depleted during 8 days.
  Interventions: Other: Beetroot juice NO3 depleted

INTERVENTIONS:
Dietary Supplement: Beetroot juice rich in nitrate — The participant will intake beetroot juice rich in NO3 (400mg) during 8-days. On the eighth day of the intervention, 2 hours after intake the last bottle of juice, the participants will return to the laboratory for the performance tests evaluation. Before crossover protocol a 7-day washout interval will be given for the purification of the compounds provided by the protocols.
  Arms: Experimental (Beetroot juice NO3)
Other: Beetroot juice NO3 depleted — The participant will intake beetroot juice depleted in NO3. On the eighth day of the intervention, 2 hours after intake the last bottle of juice, the participants will to the laboratory for the performance tests evaluation. Before crossover protocol a 7-day washout interval will be given for the purification of the compounds provided by the protocols.
  Arms: Placebo (Beetroot juice without NO3)

SUMMARY:
Through a randomized, crossover, triple-blind, placebo-controlled clinical trial, 15 physically inactive hypertensive women will participate a 8-day trial, each with two intervention protocols: 1) placebo and 2) beetroot; in which will ingest beet juice with or without NO3 in its composition with a 8-day washout interval.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 65 years old
* Physically inactive
* Postmenopausal diagnosis (amenorrhea for 12 months or more);

Exclusion Criteria:

* Smoking
* Cardiac failure
* Previous history of acute myocardial infarction and/or stroke;
* Allergy or intolerance to nitrate, gluten, or milk;

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-08-20 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength test (kgf) | up to 2 years

SECONDARY OUTCOMES:
Six minute walk test (distance in meters) | up to 2 years
Arm curl test (repetitions) | up to 2 years
Sit-to-stand test (repetitions) | up to 2 years
8-foot up and go test (seconds) | up to 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Cicero Jonas Rodrigues Benjamim, Ribeirão Preto, São Paulo
  - EEFERP - USP / Laboratório de Fisiologia do Exercício e Metabolismo, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Benjamim CJR, Lopes da Silva LS, da Silva Goncalves L, Tasinafo Junior MF, Spellanzon B, Rebelo MA, Tanus-Santos JE, Bueno Junior CR. The effects of dietary nitrate ingestion on physical performance tests in 50-65 years old postmenopausal women: A pilot randomized, double-blind, placebo-controlled, and crossover study. Clin Nutr. 2024 Jul;43(7):1642-1646. doi: 10.1016/j.clnu.2024.05.031. Epub 2024 May 22. PMID 38805867